CLINICAL TRIAL: NCT00406081
Title: Immune Response to Varicella Vaccination in Subjects With Atopic Dermatitis Compared to Nonatopic Controls (VAR 05)
Brief Title: Immune Response to Varicella Vaccination in Children With Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT ADVN VAR 05; Contract No. HHSN266200400029C
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Blood collected for endpoint measurements.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants with AD: Children with AD who received the chicken pox vaccine 2 to 16 weeks prior to the study visit (including a group of AD subjects with eczema herpeticum)
- Nonatopic controls: Children without AD who received the chicken pox vaccine 2 to 16 weeks prior to the study visit

SUMMARY:
Atopic dermatitis (AD) causes people to be susceptible to skin infection and inflammations. The purpose of this study is to determine the immune response to chicken pox vaccine in children with or without AD who received the vaccine 2 to 16 weeks prior to the study visit.

DETAILED DESCRIPTION:
AD is a chronic inflammatory skin disorder characterized by recurrent viral skin infections. Children with AD given the smallpox vaccine could develop a life-threatening condition known as eczema vaccinatum. This immune response is not currently understood. The purpose of this study is to understand the immune response to a viral vaccine in children with AD. This will be accomplished by studying immune response to the chicken pox vaccine in children with AD in comparison to those without AD.

This study will consist of one study visit occurring about 2 to 16 weeks after the child received the chicken pox vaccination. During this visit, physical and skin exams will occur. Personal and family medical histories and blood collection will also occur. The chicken pox vaccine will not be given as a part of this study. Subjects will receive the results of radioallergosorbent (RAST) testing that will tell if they are allergic to some common items (e.g., mold, grass).

ELIGIBILITY:
Inclusion Criteria:

* Parent/guardian has signed informed consent
* Male or female of any race or ethnicity
* 12 to 36 months of age, inclusive
* Healthy subjects with no systemic disorders and subjects with moderate to severe AD including a group of subjects with ADEH+
* Previously vaccinated for varicella by a physician 3 weeks prior to the Study Visit (subjects receiving the vaccine 2-16 weeks prior will also be accepted)

Exclusion Criteria:

* History of infection with chicken pox
* Oral, intravenous, or intramuscular corticosteroids within 30 days prior to chicken pox immunization
* Asthmatics receiving more than 500 micrograms per day of inhaled budesonide or more than 220 micrograms per day of inhaled fluticasone
* Antiherpes antiviral agents within 7 days prior to immunization
* Suspected immune deficiency or family history of primary immunodeficiency
* History of or active cancer
* Active untreated tuberculosis (TB)
* Respiratory illness at the time of chicken pox vaccination
* Receipt of blood products or chicken pox zoster immune globulin within the last 5 months prior to study entry

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with or without AD who received the chicken pox vaccine including a group of AD subjects with eczema herpeticum (ADEH+)
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2005-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Cell-mediated immune responses as assessed by measurement of numbers of VZV specific T cells. | 36 months

SECONDARY OUTCOMES:
To determine if children with AD have VZV-specific humoral responses to varicella vaccination that differ from those of nonatopic controls. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Schneider, MD, Study Chair — Boston Children's Hospital; Donald Y. Leung, MD, PhD, Principal Investigator — National Jewish Health
Locations (2):
- United States (2):
  - National Jewish Health, Denver, Colorado
  - Children's Hospital Boston, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Result] Schneider L, Weinberg A, Boguniewicz M, Taylor P, Oettgen H, Heughan L, Zaccaro D, Armstrong B, Holliday A, Leung DY. Immune response to varicella vaccine in children with atopic dermatitis compared with nonatopic controls. J Allergy Clin Immunol. 2010 Dec;126(6):1306-7.e2. doi: 10.1016/j.jaci.2010.08.010. PMID 20889193
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY2 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY2 — ImmPort study identifier is SDY2.
- Available data/document: Study Protocol: SDY2 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY2 — ImmPort study identifier is SDY2.
- Available data/document: Study design, -schedule of events, -demographics, -adverse events, -interventions, -files: SDY2 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY2 — ImmPort study identifier is SDY2.